CLINICAL TRIAL: NCT06392438
Title: Combination of 0.09% Cyclosporine and Intense Pulsed Light (IPL) Therapy for the Treatment of Dry Eye Disease in Symptomatic Contact Lens Wearers: a Sham-Controlled Randomized Clinical Trial
Brief Title: Cyclosporine and Intense Pulsed Light for Dry Eye in Contact Lens Users
Acronym: CycliP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Patrick Boissy, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-5200
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Dry Eye; Contact Lens Complication
Keywords: Contact Lens Discomfort; Intense Pulsed Light; Cyclosporine
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins; Intense Pulsed Light Therapy

STUDY DESIGN:
Intervention Model Description: This study is a randomized, sham controlled clinical trial. It consists of two treatments, one of which is applied to all the participants (cyclosporine). and the second one, for which participants are randomized in either the IPL group (experimental) or the IPL-sham group (control). Data collection is a pre-post model, with data being collected at baseline, during the trial (mid-study) and after the treatments. Data analysis is in intent-to-treat.
Who Masked: Participant
Masking Description: Participants will be unaware of their allocation in either the experimental group (IPL) or the control group (sham-IPL). Due to the nature of the treatment, it was not possible to mask the researcher that is performing the IPL treatment. Meibography score and conjunctival staining (requiring clinical judgment) will be analyzed by assessors that are masked (from images captured by a non-masked investigator).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IPL group (Experimental): Participants will receive 0.09% cyclosporine drops dosed at bid for 16 weeks. Participants receive 3 IPL sessions at 3-weeks interval in the last 2 months of the study. IPL treatments will be given with Lumenis M22 with a 590nm filter, pulse duration of 6-50ms (3 pulses/trigger) and fluence will be determined after determining the skin type (Fitzpatrick scale) of the participant.
  Interventions: Drug: CycloSPORINE Ophthalmic; Procedure: Intense Pulsed Light
- Sham-IPL group (Sham Comparator): Participants will receive 0.09% cyclosporine drops dosed at bid for 16 weeks. Participants receive 3 IPL sessions at 3-weeks interval in the last 2 months of the study. IPL treatments will be given with Lumenis M22 with a 590nm filter, pulse duration of 6-50ms (3 pulses/trigger) and fluence will be determined set at 10 J/cm2. A plastic filter will recover the IPL prism, preventing the light to reach the skin of the participant.
  Interventions: Drug: CycloSPORINE Ophthalmic; Procedure: Sham Intense Pulse Light

INTERVENTIONS:
Drug: CycloSPORINE Ophthalmic — Unidose of Cequa provided without charge to the participant. 1 drop in each eye morning and evening.
  Other Names: Cequa
Procedure: Intense Pulsed Light — Appropriate eye patches and IPL gel will be applied. 15 triggers per passage will be applied from the right temple to the left temple (7 shots from the right temple to the right nose wing, 1 on the nose bridge and 7 shots from the left nose wing to the left temple). 2 passage/session will be applied.
  Other Names: IPL M22 Lumenis
  Arms: IPL group
Procedure: Sham Intense Pulse Light — Appropriate eye patches and IPL gel will be applied. 15 triggers per passage will be applied with the plastic blocker mounted on the IPL prism from the right temple to the left temple (7 shots from the right temple to the right nose wing, 1 on the nose bridge and 7 shots from the left nose wing to the left temple). 2 passage/session will be applied.
  Other Names: Sham-IPL M22 Lumenis
  Arms: Sham-IPL group

SUMMARY:
In this study, two treatments typically used for dry eye disease will be tried for contact lens users to see if their symptoms when they use their contact lenses get better. Cyclosporine is a drop that is used for long-term management of the inflammation and Intense pulsed light (IPL) is a treatment done in a clinic to improve the health of the eyelid glands. The main question in this study is:

Does the combined treatment of cyclosporine and IPL improve the symptoms and the dry eye signs of contact lens wearers?

All the participants will receive the cyclosporine drops for 4 months twice a day. The research team will split the group of participants in two, half receiving the real IPL treatment and half receiving a sham IPL treatment during the last two months of the study. This will allow to compare the two groups to see how IPL helped. The dry eye tests will be done at the start of the study, after two months and after 4 months. The tests will include a dry eye symptoms questionnaire, measures on the tears, the structures of the front of the eye and the eyelids.

DETAILED DESCRIPTION:
Dry eye disease is a complex and multifactorial pathology in which inflammation and changes to the tear film (instability and hyperosmolarity) play important roles. Dry eye disease is very common, with an estimated global prevalence of 11.59% although other analyses conclude to 50% of some populations suffering from dry eye. The condition has been traditionally classified in two subtypes: aqueous tear deficiency (secondary to a deficit of production by the lacrimal gland) and evaporative disease (secondary to a deficit of the lipid layer of the tear film), but when the condition progresses, almost all patients present characteristics of both subtypes. Meibomian gland dysfunction (MGD) is one of the conditions that is most frequently associated with dry eye disease and leads to evaporative dry eye and alterations of the ocular surface. The prevalence of MGD has been recently established between 21.2% and 29.5% in subjects of African and Caucasian race and higher among Arabs, Hispanics, and Asians. Many risk factors exist for dry eye disease and MGD, including age and usage of contact lens. Soft contact lenses (SCL) are used by hundreds of millions for visual correction. The wear of SCL, however, has the potential to create or worsen dry eye signs and symptoms. A comparative study has found that 39% of North-American wearers can be categorized as symptomatic of contact lens dry eye and the proportion of uncomfortable users increases with age. SCL wear can increase evaporative dry eye by weakening the lipid layer, which leads to decreased stability of the tear film and increased evaporation. It also contributes to aqueous dry eye etiology by reducing the tear volume. The wear of SCL has also been shown to have a damaging effect on meibomian glands and, in some cases, on the conjunctival goblet cells .

Arguments also support the role of SCL in the inflammation of the ocular surface, even in asymptomatic patients. Thus, dry eye disease associated with SCL wear is a complex condition that implies different mechanisms.

Cyclosporine A is a peptide produced by a fungus that has been used systemically for decades for its potent immunomodulatory effects. Usage for dry eye disease in a topical 0.05% oil-based formulation has been common since the early 2000s. On the ocular surface, cyclosporine acts by inhibiting calcineurin, which subsequently blocks the activation of T cells and prevents the release of cytokines, therefore reducing inflammation. It has been shown to increase tear volume, goblet cell density and to reduce surface staining as well as symptoms in dry eye patients. Divergent results have been observed on contact lens wearers, although one study has found an amplified effect on contact lens wearers symptomatic of dry eye when combining essential fatty acid supplements with topical cyclosporine. Despite having been shown useful in the management of dry eye disease, the oil-based formulation is considered having a low bioavailability. A new cyclosporine eyedrop has been approved in Canada and the USA in the recent past years and is based on nanomicelle technology with a concentration of 0.09%. This nano-micellar formulation could be more effective in delivering the cyclosporine to the tissues and have been shown to reduce ocular surface staining, to increase tear volume, and to be safe. Adverse events that are known to this product are mild, such as transient pain at instillation for about 23% of patients.

Intense pulsed light (IPL) is a therapeutic process that has been used for many years in dermatology and esthetics. The noncoherent pulses of light produce photo-biochemical effects and, in the treatment of dry eye disease, the application on the skin around the orbit to produces these effects on the meibomian glands and their surrounding tissue. The mechanisms by which IPL improves signs and symptoms of dry eye are not fully understood, but the melting of the meibum, the clogging of telangiectatic inflammatory vessels, the reduction of epithelial turnover, the improvement in the collagen synthesis, a mitochondrial activity enhancement (photo modulation), and the destruction of parasitic and bacterial species are the main theoretical explanations. IPL has been shown to be an effective therapeutic option to manage MGD.

Dozens of studies have shown that IPL reduces dry eye symptoms, increases tear break-up time, improves the secreting function of the glands as well as the quality of the meibum and reduces corneal staining. IPL is often combined with meibomian gland expression to maximize the therapeutic effects; however, controlled studies have shown that IPL is largely responsible of these effects and that it is the core mechanism of this combination. Two studies have observed the effect of IPL on SCL users, with the conclusion that it is an effective treatment for this population. IPL is considered to be a safe treatment.

Since SCL have been linked to both aqueous and evaporative etiologies or dry eye, this research project aims to study the effect of combining these two treatments to target the entirety of the tear film, believed to be essential to comfortable SCL wear. This study will be a randomized clinical trial that contains two interventions: the 0.09% cyclosporine eyedrops (Cequa) and IPL treatment. The main objective of this study is to establish if the treatment of contact lens related dry eyes by the combination of 0.09% cyclosporine for 16 weeks and a standard IPL treatment (3 sessions) is more effective in relieving dry eye symptoms when compared to 0.09% cyclosporine for 16 weeks with a sham IPL treatment (3 sessions). The secondary objectives are to compare the effects of each treatment combination (0.09% cyclosporine+IPL vs 0.09% cyclosporine+sham) on signs of dry eye, to explore the effects of cyclosporine 0.09% drops alone on contact lens wearers and to assess the security profile of these interventions on SCL wearers.

Based on prior data from the f-CLDEQ-8 validation study, a major study on the cyclosporine nanomicelle formulation and the first clinical trial on IPL for contact lens wearers, a sample size of 44 participants (22/group) was calculated to be necessary to detect a significant difference between the groups. 44 participants will thus be recruited from a primary care optometric clinic and nearby clinics. Participation to the study will require 5 visits from the participants. The first visit will be a collection of data and the dispensing of the 0.09% cyclosporine drops. 8 weeks later, the participants will present for their 2nd visit, during which data will be collected once again and participants will be randomized to either the treatment or the sham group and will receive their first treatment (IPL or sham accordingly to the assignation). The 2 following visits, 3 weeks apart, will be for the 2 last IPL/sham treatments. A final visit will be for data collection 2 weeks after the last IPL/sham treatment. Participants will take 0.09% cyclosporine for the whole 16 weeks.

A bilateral t-test for independent samples will be used to compare the difference in change on the f-CLDEQ-8 between groups on the 16 weeks interval. Concerning the dry eye signs, statistical treatment will be made to account for inter-eye correlation. Continuous variables will be analyzed using a multi-level model to assess the difference in change between groups on the 16 weeks interval. Discrete variable will be analyzed using a general linear model (GLM) for the same comparison. Data will be handled in an intent-to-treat way.

ELIGIBILITY:
Inclusion Criteria:

* Soft silicone-hydrogel contact lens wearers
* Monthly, 2-weeks, opr daily replacement schedule of contact lens
* Minimum wear of contact lens for 1 day/week and 4 hours consecutive
* f-CLDEQ-8 score ≥ 12

Exclusion Criteria:

* Past usage of cyclosporine 0.09% (Cequa)
* Use of another ophthalmic cyclosporine drop in the past 6 months
* Known intolerance to cyclosporine
* Pregnancy or breastfeeding (or planned pregnancy in the duration study)
* History of ocular herpes simplex infection
* Active ocular infectious condition
* Usage of photosensitizing medication
* Epilepsy
* History of skin cancer in the IPL treatment zone
* Tattoo/pigmented lesion/keloid scars in the IPL treatment zone
* Refractive surgery in the past 12 months
* In-clinic thermal pulsation eyelid treatment in the past 12 months
* Usage of glaucoma drops
* Regular continuous wear of contact lenses (including sleep)
* Excessive movement or decentration of the contact lenses (assessed at first visit)
* Giant papillary conjunctivitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Contact lens dry eye symptoms | Measured at each visit (Baseline, week 8, week 11, week 14 and week 16)
  f-CLDEQ-8 questionnaire (French version of the Contact Lens Dry Eye Questionnaire - 8). Scores possible are from 1 to 37; higher score means more symptoms and worse dry eye

SECONDARY OUTCOMES:
Global rating scale of change | Tuesday and Saturday of every week for 16 consecutive weeks (while participating in the study)
  Rating 0-100 of perceived comfort during contact lens wear in the past days; question sent by platform of ecological momentary assessment REDCap
Average number of hours spent wearing contact lenses | Tuesday and Saturday of every week for 16 consecutive weeks (while participating in the study))
  Question sent by platform of ecological momentary assessment REDCap
Artificial tear usage while wearing contact lenses | Tuesday and Saturday of every week for 16 consecutive weeks (while participating in the study)
  Question sent by platform of ecological momentary assessment REDCap
Non-invasive tear break-up time over contact lenses (pre-lens tear film) | Baseline, week 8, and week 16
  Measured with the TFSQ NIBUT of the Medmont corneal topographer
Non-invasive tear break-up time (natural tear film) | Baseline, week 8, and week 16
  Measured with the TFSQ NIBUT of the Medmont E300 corneal topographer
Tear break-up time | Baseline, week 8, and week 16
  Average of 3 readings with fluorescein and observation through a slit lamp using cobalt and yellow filter
Corneal staining score | Baseline, week 8, and week 16
  Pictures of the cornea taken through an anterior segment imagery system (mounted on slit lamp) after fluorescein instillation. Pictures analyzed by automated AOS system, which counts the exact number of corneal punctate lesions
Conjunctival staining score | Baseline, week 8, and week 16
  Pictures of the nasal and temporal conjunctiva taken through an anterior segment imagery system (mounted on slit lamp) after lissamine green instillation. Pictures analyzed by masked experienced rater and graded using Efron grading scale (grade 0 to 4, a higher score meaning worse condition)
Tear meniscus height (with contact lens in place) | Baseline, week 8, and week 16
  Measured at the inferior meniscus with the Myah (Topcon) automated function before contact lens removal
Tear osmolarity (with contact lens in place) | Baseline, week 8, and week 16
  Measured on inferior palpebral conjunctiva with the iPen (i-Med) before contact lens removal
Meibomian gland atrophy | Baseline and week 16
  Meibography scans performed on all 4 eyelids with the Lipiscan (Johnson & Johnson) and sent to masked experienced rater for rating using the Meiboscore (Pult)
Adverse effects | Week 8, week 11, week 14, and week 16
  Measured with home questionnaire containing 16 questions on adverse effects from both interventions
Distance visual acuity | Measured at each visit (Baseline, week 8, week 11, week 14 and week 16)
  Variable measured for safety assessment. Snellen chart used with current correction (contact lens or glasses)
Intraocular pressure | Measured at each visit (Baseline, week 8, week 11, week 14 and week 16)
  Variable measured for safety assessment. Non-contact airpuff tonometer (Nidek RKT-7700)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Boissy, PhD, Study Chair — Professor University of Sherbrooke; Langis Michaud, OD, MSc, Study Director — Professor University of Montreal; Eric Lortie-Milner, OD, Principal Investigator — PhD candidate University of Sherbrooke
Locations (1):
- Opto-Réseau Sherbrooke Est, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Raw data and individual participant data (denominalized) will be available upon reasonable demand to the research team.
  Protocol article will be submitted for publication
Supporting Information: Study Protocol, SAP
Time Frame: Any time after publication of the results from this trial
Access Criteria: Verified scholar; clearly stated motive and need for the data; plan to securely store the data.

REFERENCES:
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Papas EB. The global prevalence of dry eye disease: A Bayesian view. Ophthalmic Physiol Opt. 2021 Nov;41(6):1254-1266. doi: 10.1111/opo.12888. Epub 2021 Sep 21. PMID 34545606
- [Background] Stapleton F, Alves M, Bunya VY, Jalbert I, Lekhanont K, Malet F, Na KS, Schaumberg D, Uchino M, Vehof J, Viso E, Vitale S, Jones L. TFOS DEWS II Epidemiology Report. Ocul Surf. 2017 Jul;15(3):334-365. doi: 10.1016/j.jtos.2017.05.003. Epub 2017 Jul 20. PMID 28736337
- [Background] Rouen PA, White ML. Dry Eye Disease: Prevalence, Assessment, and Management. Home Healthc Now. 2018 Mar/Apr;36(2):74-83. doi: 10.1097/NHH.0000000000000652. PMID 29498987
- [Background] Chhadva P, Goldhardt R, Galor A. Meibomian Gland Disease: The Role of Gland Dysfunction in Dry Eye Disease. Ophthalmology. 2017 Nov;124(11S):S20-S26. doi: 10.1016/j.ophtha.2017.05.031. PMID 29055358
- [Background] Hassanzadeh S, Varmaghani M, Zarei-Ghanavati S, Heravian Shandiz J, Azimi Khorasani A. Global Prevalence of Meibomian Gland Dysfunction: A Systematic Review and Meta-Analysis. Ocul Immunol Inflamm. 2021 Jan 2;29(1):66-75. doi: 10.1080/09273948.2020.1755441. Epub 2020 Jun 26. PMID 32589483
- [Background] Schaumberg DA, Nichols JJ, Papas EB, Tong L, Uchino M, Nichols KK. The international workshop on meibomian gland dysfunction: report of the subcommittee on the epidemiology of, and associated risk factors for, MGD. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1994-2005. doi: 10.1167/iovs.10-6997e. Print 2011 Mar. No abstract available. PMID 21450917
- [Background] Gomes JAP, Azar DT, Baudouin C, Efron N, Hirayama M, Horwath-Winter J, Kim T, Mehta JS, Messmer EM, Pepose JS, Sangwan VS, Weiner AL, Wilson SE, Wolffsohn JS. TFOS DEWS II iatrogenic report. Ocul Surf. 2017 Jul;15(3):511-538. doi: 10.1016/j.jtos.2017.05.004. Epub 2017 Jul 20. PMID 28736341
- [Background] Dumbleton K, Caffery B, Dogru M, Hickson-Curran S, Kern J, Kojima T, Morgan PB, Purslow C, Robertson DM, Nelson JD; members of the TFOS International Workshop on Contact Lens Discomfort. The TFOS International Workshop on Contact Lens Discomfort: report of the subcommittee on epidemiology. Invest Ophthalmol Vis Sci. 2013 Oct 18;54(11):TFOS20-36. doi: 10.1167/iovs.13-13125. No abstract available. PMID 24058130
- [Background] Koh S. Contact Lens Wear and Dry Eye: Beyond the Known. Asia Pac J Ophthalmol (Phila). 2020 Dec;9(6):498-504. doi: 10.1097/APO.0000000000000329. PMID 33284229
- [Background] Chalmers RL, Young G, Kern J, Napier L, Hunt C. Soft Contact Lens-Related Symptoms in North America and the United Kingdom. Optom Vis Sci. 2016 Aug;93(8):836-47. doi: 10.1097/OPX.0000000000000927. PMID 27391535
- [Background] Sulley A, Young G, Hunt C, McCready S, Targett MT, Craven R. Retention Rates in New Contact Lens Wearers. Eye Contact Lens. 2018 Sep;44 Suppl 1:S273-S282. doi: 10.1097/ICL.0000000000000402. PMID 28617731
- [Background] Bron AJ, de Paiva CS, Chauhan SK, Bonini S, Gabison EE, Jain S, Knop E, Markoulli M, Ogawa Y, Perez V, Uchino Y, Yokoi N, Zoukhri D, Sullivan DA. TFOS DEWS II pathophysiology report. Ocul Surf. 2017 Jul;15(3):438-510. doi: 10.1016/j.jtos.2017.05.011. Epub 2017 Jul 20. PMID 28736340
- [Background] Guillon M, Maissa C. Contact lens wear affects tear film evaporation. Eye Contact Lens. 2008 Nov;34(6):326-30. doi: 10.1097/ICL.0b013e31818c5d00. PMID 18997542
- [Background] Nichols JJ, Sinnott LT. Tear film, contact lens, and patient-related factors associated with contact lens-related dry eye. Invest Ophthalmol Vis Sci. 2006 Apr;47(4):1319-28. doi: 10.1167/iovs.05-1392. PMID 16565363
- [Background] Alghamdi WM, Markoulli M, Holden BA, Papas EB. Impact of duration of contact lens wear on the structure and function of the meibomian glands. Ophthalmic Physiol Opt. 2016 Mar;36(2):120-31. doi: 10.1111/opo.12278. PMID 26890701
- [Background] Ucakhan O, Arslanturk-Eren M. The Role of Soft Contact Lens Wear on Meibomian Gland Morphology and Function. Eye Contact Lens. 2019 Sep;45(5):292-300. doi: 10.1097/ICL.0000000000000572. PMID 30608243
- [Background] Insua Pereira E, Sampaio AP, Lira M. Effects of contact lens wear on tear inflammatory biomarkers. Cont Lens Anterior Eye. 2022 Oct;45(5):101600. doi: 10.1016/j.clae.2022.101600. Epub 2022 Apr 21. PMID 35466056
- [Background] Alzahrani Y, Colorado LH, Pritchard N, Efron N. Longitudinal changes in Langerhans cell density of the cornea and conjunctiva in contact lens-induced dry eye. Clin Exp Optom. 2017 Jan;100(1):33-40. doi: 10.1111/cxo.12399. Epub 2016 Jun 28. PMID 27353750
- [Background] Efron N. Contact lens wear is intrinsically inflammatory. Clin Exp Optom. 2017 Jan;100(1):3-19. doi: 10.1111/cxo.12487. Epub 2016 Nov 2. PMID 27806431
- [Background] Periman LM, Mah FS, Karpecki PM. A Review of the Mechanism of Action of Cyclosporine A: The Role of Cyclosporine A in Dry Eye Disease and Recent Formulation Developments. Clin Ophthalmol. 2020 Dec 2;14:4187-4200. doi: 10.2147/OPTH.S279051. eCollection 2020. PMID 33299295
- [Background] Wan KH, Chen LJ, Young AL. Efficacy and Safety of Topical 0.05% Cyclosporine Eye Drops in the Treatment of Dry Eye Syndrome: A Systematic Review and Meta-analysis. Ocul Surf. 2015 Jul;13(3):213-25. doi: 10.1016/j.jtos.2014.12.006. Epub 2015 Apr 11. PMID 26045239
- [Background] Rao SN. Topical cyclosporine 0.05% for the prevention of dry eye disease progression. J Ocul Pharmacol Ther. 2010 Apr;26(2):157-64. doi: 10.1089/jop.2009.0091. PMID 20415623
- [Background] Chen M, Gong L, Sun X, Xie H, Zhang Y, Zou L, Qu J, Li Y, He J. A comparison of cyclosporine 0.05% ophthalmic emulsion versus vehicle in Chinese patients with moderate to severe dry eye disease: an eight-week, multicenter, randomized, double-blind, parallel-group trial. J Ocul Pharmacol Ther. 2010 Aug;26(4):361-6. doi: 10.1089/jop.2009.0145. PMID 20698799
- [Background] Prabhasawat P, Tesavibul N, Mahawong W. A randomized double-masked study of 0.05% cyclosporine ophthalmic emulsion in the treatment of meibomian gland dysfunction. Cornea. 2012 Dec;31(12):1386-93. doi: 10.1097/ICO.0b013e31823cc098. PMID 23135530
- [Background] Chen D, Zhang S, Bian A, Hong J, Deng Y, Zhang M, Chen W, Shao Y, Zhao J. Efficacy and safety of 0.05% cyclosporine ophthalmic emulsion in treatment of Chinese patients with moderate to severe dry eye disease: A 12-week, multicenter, randomized, double-masked, placebo-controlled phase III clinical study. Medicine (Baltimore). 2019 Aug;98(31):e16710. doi: 10.1097/MD.0000000000016710. PMID 31374063
- [Background] Hom MM. Use of cyclosporine 0.05% ophthalmic emulsion for contact lens-intolerant patients. Eye Contact Lens. 2006 Mar;32(2):109-11. doi: 10.1097/01.icl.0000175651.30487.58. PMID 16538135
- [Background] Willen CM, McGwin G, Liu B, Owsley C, Rosenstiel C. Efficacy of cyclosporine 0.05% ophthalmic emulsion in contact lens wearers with dry eyes. Eye Contact Lens. 2008 Jan;34(1):43-5. doi: 10.1097/ICL.0b013e3180676d44. PMID 18180683
- [Background] Wang L, Chen X, Hao J, Yang L. Proper balance of omega-3 and omega-6 fatty acid supplements with topical cyclosporine attenuated contact lens-related dry eye syndrome. Inflammopharmacology. 2016 Dec;24(6):389-396. doi: 10.1007/s10787-016-0291-2. Epub 2016 Oct 20. PMID 27766505
- [Background] Jerkins GW, Pattar GR, Kannarr SR. A Review of Topical Cyclosporine A Formulations-A Disease-Modifying Agent for Keratoconjunctivitis Sicca. Clin Ophthalmol. 2020 Feb 20;14:481-489. doi: 10.2147/OPTH.S228070. eCollection 2020. PMID 32109984
- [Background] Mandal A, Gote V, Pal D, Ogundele A, Mitra AK. Ocular Pharmacokinetics of a Topical Ophthalmic Nanomicellar Solution of Cyclosporine (Cequa(R)) for Dry Eye Disease. Pharm Res. 2019 Jan 7;36(2):36. doi: 10.1007/s11095-018-2556-5. PMID 30617777
- [Background] Weiss SL, Kramer WG. Ocular Distribution of Cyclosporine Following Topical Administration of OTX-101 in New Zealand White Rabbits. J Ocul Pharmacol Ther. 2019 Sep;35(7):395-402. doi: 10.1089/jop.2018.0106. Epub 2019 Aug 6. PMID 31355703
- [Background] Malhotra R, Devries DK, Luchs J, Kabat A, Schechter BA, Shen Lee B, Shettle L, Smyth-Medina R, Ogundele A, Darby C, Bacharach J, Karpecki P. Effect of OTX-101, a Novel Nanomicellar Formulation of Cyclosporine A, on Corneal Staining in Patients With Keratoconjunctivitis Sicca: A Pooled Analysis of Phase 2b/3 and Phase 3 Studies. Cornea. 2019 Oct;38(10):1259-1265. doi: 10.1097/ICO.0000000000001989. PMID 31306284
- [Background] Smyth-Medina R, Johnston J, Devries DK, Jasper A, Kannarr SR, Schechter BA, Shen Lee B, Varghese G, Ogundele A, Darby CH, Karpecki P, Luchs J. Effect of OTX-101, a Novel Nanomicellar Formulation of Cyclosporine A, on Conjunctival Staining in Patients with Keratoconjunctivitis Sicca: A Pooled Analysis of Phase 2b/3 and 3 Clinical Trials. J Ocul Pharmacol Ther. 2019 Sep;35(7):388-394. doi: 10.1089/jop.2018.0154. Epub 2019 Aug 2. PMID 31373837
- [Background] Sheppard J, Kannarr S, Luchs J, Malhotra R, Justice A, Ogundele A, Darby C, Bacharach J. Efficacy and Safety of OTX-101, a Novel Nanomicellar Formulation of Cyclosporine A, for the Treatment of Keratoconjunctivitis Sicca: Pooled Analysis of a Phase 2b/3 and Phase 3 Study. Eye Contact Lens. 2020 Jan;46 Suppl 1:S14-S19. doi: 10.1097/ICL.0000000000000636. PMID 31361655
- [Background] Toyos M, Gupta PK, Mitchell B, Karpecki P. The Effect of OTX-101 on Tear Production in Patients with Severe Tear-deficient Dry Eye Disease: A Pooled Analysis of Phase 2b/3 and Phase 3 Studies. Curr Eye Res. 2022 Feb;47(2):220-224. doi: 10.1080/02713683.2021.1966477. Epub 2021 Aug 29. PMID 34459350
- [Background] Sheppard J, Bergmann M, Schechter BA, Luchs J, Ogundele A, Karpecki P. Phase 3 Efficacy (Worse-Eye Analysis) and Long-Term Safety Evaluation of OTX-101 in Patients with Keratoconjunctivitis Sicca. Clin Ophthalmol. 2021 Jan 12;15:129-140. doi: 10.2147/OPTH.S279364. eCollection 2021. PMID 33469259
- [Background] Raulin C, Greve B, Grema H. IPL technology: a review. Lasers Surg Med. 2003;32(2):78-87. doi: 10.1002/lsm.10145. PMID 12561039
- [Background] Rennick S, Adcock L. Intense Pulsed Light Therapy for Meibomian Gland Dysfunction: A Review of Clinical Effectiveness and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2018 Feb 8. Available from http://www.ncbi.nlm.nih.gov/books/NBK531789/ PMID 30307727
- [Background] Dell SJ. Intense pulsed light for evaporative dry eye disease. Clin Ophthalmol. 2017 Jun 20;11:1167-1173. doi: 10.2147/OPTH.S139894. eCollection 2017. PMID 28790801
- [Background] Giannaccare G, Taroni L, Senni C, Scorcia V. Intense Pulsed Light Therapy In The Treatment Of Meibomian Gland Dysfunction: Current Perspectives. Clin Optom (Auckl). 2019 Oct 17;11:113-126. doi: 10.2147/OPTO.S217639. eCollection 2019. PMID 31802961
- [Background] Suwal A, Hao JL, Zhou DD, Liu XF, Suwal R, Lu CW. Use of Intense Pulsed Light to Mitigate Meibomian Gland Dysfunction for Dry Eye Disease. Int J Med Sci. 2020 Jun 1;17(10):1385-1392. doi: 10.7150/ijms.44288. eCollection 2020. PMID 32624695
- [Background] Craig JP, Chen YH, Turnbull PR. Prospective trial of intense pulsed light for the treatment of meibomian gland dysfunction. Invest Ophthalmol Vis Sci. 2015 Feb 12;56(3):1965-70. doi: 10.1167/iovs.14-15764. PMID 25678687
- [Background] Piyacomn Y, Kasetsuwan N, Reinprayoon U, Satitpitakul V, Tesapirat L. Efficacy and Safety of Intense Pulsed Light in Patients With Meibomian Gland Dysfunction-A Randomized, Double-Masked, Sham-Controlled Clinical Trial. Cornea. 2020 Mar;39(3):325-332. doi: 10.1097/ICO.0000000000002204. PMID 31764289
- [Background] Xue AL, Wang MTM, Ormonde SE, Craig JP. Randomised double-masked placebo-controlled trial of the cumulative treatment efficacy profile of intense pulsed light therapy for meibomian gland dysfunction. Ocul Surf. 2020 Apr;18(2):286-297. doi: 10.1016/j.jtos.2020.01.003. Epub 2020 Jan 30. PMID 32007523
- [Background] Toyos R, Desai NR, Toyos M, Dell SJ. Intense pulsed light improves signs and symptoms of dry eye disease due to meibomian gland dysfunction: A randomized controlled study. PLoS One. 2022 Jun 23;17(6):e0270268. doi: 10.1371/journal.pone.0270268. eCollection 2022. PMID 35737696
- [Background] Miao S, Yan R, Jia Y, Pan Z. Effect of Intense Pulsed Light Therapy in Dry Eye Disease Caused by Meibomian Gland Dysfunction: A Systematic Review and Meta-Analysis. Eye Contact Lens. 2022 Oct 1;48(10):424-429. doi: 10.1097/ICL.0000000000000934. Epub 2022 Sep 5. PMID 36044829
- [Background] Sambhi RS, Sambhi GDS, Mather R, Malvankar-Mehta MS. Intense pulsed light therapy with meibomian gland expression for dry eye disease. Can J Ophthalmol. 2020 Jun;55(3):189-198. doi: 10.1016/j.jcjo.2019.11.009. Epub 2020 Jan 13. PMID 31941589
- [Background] Arita R, Fukuoka S, Morishige N. Therapeutic efficacy of intense pulsed light in patients with refractory meibomian gland dysfunction. Ocul Surf. 2019 Jan;17(1):104-110. doi: 10.1016/j.jtos.2018.11.004. Epub 2018 Nov 13. PMID 30445177
- [Background] Rong B, Tang Y, Tu P, Liu R, Qiao J, Song W, Toyos R, Yan X. Intense Pulsed Light Applied Directly on Eyelids Combined with Meibomian Gland Expression to Treat Meibomian Gland Dysfunction. Photomed Laser Surg. 2018 Jun;36(6):326-332. doi: 10.1089/pho.2017.4402. Epub 2018 Apr 24. PMID 29688838
- [Background] Shin KY, Lim DH, Moon CH, Kim BJ, Chung TY. Intense pulsed light plus meibomian gland expression versus intense pulsed light alone for meibomian gland dysfunction: A randomized crossover study. PLoS One. 2021 Mar 4;16(3):e0246245. doi: 10.1371/journal.pone.0246245. eCollection 2021. PMID 33662017
- [Background] Yang L, Pazo EE, Zhang Q, Wu Y, Song Y, Qin G, Zhang H, Li J, Xu L, He W. Treatment of contact lens related dry eye with intense pulsed light. Cont Lens Anterior Eye. 2022 Apr;45(2):101449. doi: 10.1016/j.clae.2021.101449. Epub 2021 Apr 28. PMID 33933353
- [Background] Xu L, Wu Y, Song Y, Zhang Q, Qin G, Yang L, Ma J, Palme C, Moore JE, Pazo EE, He W. Comparison Between Heated Eye Mask and Intense Pulsed Light Treatment for Contact Lens-Related Dry Eye. Photobiomodul Photomed Laser Surg. 2022 Mar;40(3):189-197. doi: 10.1089/photob.2021.0094. PMID 35298282
- [Background] Yan S, Wu Y. Efficacy and safety of Intense pulsed light therapy for dry eye caused by meibomian gland dysfunction: a randomised trial. Ann Palliat Med. 2021 Jul;10(7):7857-7865. doi: 10.21037/apm-21-1303. PMID 34353073
- [Background] Lortie-Milner E, Boily L, Michaud L, Quesnel NM, Simard P, Milner V, Boissy P. Translation and validation of the contact lens dry eye questionnaire 8 (CLDEQ-8) in Canadian French. Cont Lens Anterior Eye. 2023 Apr;46(2):101779. doi: 10.1016/j.clae.2022.101779. Epub 2022 Dec 6. PMID 36481132
- [Background] Tauber J, Schechter BA, Bacharach J, Toyos MM, Smyth-Medina R, Weiss SL, Luchs JI. A Phase II/III, randomized, double-masked, vehicle-controlled, dose-ranging study of the safety and efficacy of OTX-101 in the treatment of dry eye disease. Clin Ophthalmol. 2018 Oct 2;12:1921-1929. doi: 10.2147/OPTH.S175065. eCollection 2018. PMID 30323548
- [Background] Downie LE, Gad A, Wong CY, Gray JHV, Zeng W, Jackson DC, Vingrys AJ. Modulating Contact Lens Discomfort With Anti-Inflammatory Approaches: A Randomized Controlled Trial. Invest Ophthalmol Vis Sci. 2018 Jul 2;59(8):3755-3766. doi: 10.1167/iovs.18-24758. PMID 30046817
- [Background] Downie LE. Automated Tear Film Surface Quality Breakup Time as a Novel Clinical Marker for Tear Hyperosmolarity in Dry Eye Disease. Invest Ophthalmol Vis Sci. 2015 Nov;56(12):7260-8. doi: 10.1167/iovs.15-17772. PMID 26544794
- [Background] Walker MK, Tomiyama ES, Skidmore KV, Assaad JR, Ticak A, Richdale K. A comparison of subjective and objective conjunctival hyperaemia grading with AOS(R) Anterior software. Clin Exp Optom. 2022 Jul;105(5):494-499. doi: 10.1080/08164622.2021.1945406. Epub 2021 Jul 27. PMID 34315357
- [Background] Efron N, Morgan PB, Katsara SS. Validation of grading scales for contact lens complications. Ophthalmic Physiol Opt. 2001 Jan;21(1):17-29. PMID 11220037
- [Background] Fagehi R, Al-Bishry AB, Alanazi MA, Abusharha A, El-Hiti GA, Masmali AM. Investigation of the repeatability of tear osmolarity using an I-PEN osmolarity device. Taiwan J Ophthalmol. 2020 Dec 17;11(2):168-174. doi: 10.4103/tjo.tjo_65_20. eCollection 2021 Apr-Jun. PMID 34295623
- [Background] Pult H, Riede-Pult B. Comparison of subjective grading and objective assessment in meibography. Cont Lens Anterior Eye. 2013 Feb;36(1):22-7. doi: 10.1016/j.clae.2012.10.074. Epub 2012 Oct 27. PMID 23108007
- [Derived] Lortie-Milner E, Michaud L, Dubois MF, Boissy P. Combination of 0.09% cyclosporine and intense pulsed light (IPL) therapy for the treatment of dry eye disease in symptomatic contact lens wearers: study protocol for a sham-controlled randomized clinical trial. Trials. 2026 Feb 7. doi: 10.1186/s13063-026-09521-w. Online ahead of print. PMID 41654845

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT06392438/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT06392438/ICF_001.pdf